CLINICAL TRIAL: NCT04043585
Title: Effects of Bariatric Surgery on Non-Alcoholic Steatohepatitis
Brief Title: Bariatric Surgery on NASH
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Gubra ApS (Unknown)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, head of department, University Hospital, Gentofte, Copenhagen
Other Study IDs: EBSoNAS
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsies for histological and transcriptomic assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study investigates non-alcoholic fatty liver disease from serial liver biopsies collected from participants referred for assessment of bariatric surgery, RYGB or SG.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is an increasing health care problem closely related to obesity and has become the most common cause of chronic liver disease in developed countries. Today, bariatric surgery is the most efficient treatment of morbid obesity in terms of a rapid and sustained loss of weight. In addition, bariatric surgery is accompanied by improvement of weight-related comorbidities including features of the metabolic syndrome and possibly regression of the entire NAFLD spectrum.

The study is designed as an observational study including 40 patients referred to laparoscopic bariatric surgery (either RYGB or SG). The primary endpoint is change in NAFLD activity score (NAS) in serial liver biopsies collected from participants. Additional tests include blood samples, anthropometry measurements, Fibroscan and full body dual-energy X-ray absorptiometry (DEXA) scan performed together with each biopsy.

This unique model of serial liver biopsies in morbidly obese patients referred to bariatric surgery (RYGB or SG), combined with state-of-the-art technologies and bioinformatics, will provide important information about the effects of weight loss on NASH. The results will improve our understanding of the underlying mechanisms with the potential of identifying new potential NASH targets or diagnostic biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI≥35 kg/m2) individuals referred for bariatric surgery, either RYGB or SG
* Age between 18 and 60 years at the time of inclusion
* Evidence of potential NASH with fibrosis
* Willing to give informed consent and comply with all study procedures

Exclusion Criteria:

* Type 1 diabetes
* Alcohol consumption ≥20 g/day for women or ≥30 g/day for men over a two-year period prior to inclusion
* Clinically significant kidney function impairment or other laboratory findings at time of screening leading to the diagnosis of clinically relevant disorders
* Any physical or psychological condition that the investigator evaluates would interfere with trial participation
* Previous gastrointestinal surgery (excluding cholecystectomy and appendectomy)
* Planned elective surgery (other than bariatric surgery) during the study period with the exception of dermatosurgical, ENT (ear, nose, throat) or dental procedures not requiring general anaesthesia and/or perioperative antibiotic treatment
* Pregnancy or desire to become pregnant during the study period
* Any ongoing medication that the investigator evaluates would interfere with trial participation including anticoagulant medication, and medication that could cause NAFLD
* Contraindications to liver biopsy
* Other causes of liver disease than NAFLD, including viral hepatitis, Wilsons disease, cystic fibrosis, coeliac disease and alpha-1 antitrypsin deficiency.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30-40 patients referred to laparoscopic bariatric surgery (either RYGB or SG)
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
NAFLD activity score | 18 months
  Change in NAFLD activity score (NAS). Assessment of NAS, a standardized tool for assessment of liver histology, is often used for quantification of disease activity, allowing comparison of biopsies in clinical studies and improved reproducibility. The NAS is defined as the sum of scores for steatosis (0-3), lobular inflammation (0-3) and ballooning degeneration (0-2)

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Study Director — UGGentofte
Locations (1):
- Center for Clinical Metabolic Research, Hellerup, Denmark